CLINICAL TRIAL: NCT06102330
Title: Multicenter HomeVENT: Home Values and Experiences Navigation Track
Acronym: HomeVENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00395948; 1R01HD110414-01A1 (NIH)
Record Dates: First submitted 2023-10-19; First posted 2023-10-26 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Pediatric ALL; Respiratory Insufficiency; Communication
Keywords: chronic ventilation; decision-making
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Respiratory Insufficiency; Communication

STUDY DESIGN:
Intervention Model Description: The first half of families at each site will be enrolled in the 'usual care' arm, the second half enrolled in the 'intervention' arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): No alteration in care. Will interview families and clinicians at 1 month, and families again at 6 and 12 months
- Intervention (Experimental): Will review a web-based decision-making tool with families and simultaneously interview family regarding website topics. Will interview families and clinicians at 1 month, and families again at 6 and 12 months
  Interventions: Other: HomeVENT decision support tool

INTERVENTIONS:
Other: HomeVENT decision support tool — Web-based decision support tool that describes diverse family experiences with making decisions about pediatric chronic home ventilation
  Arms: Intervention

SUMMARY:
This is a multicenter study to test a decision-making support process for families and clinicians facing decisions about chronic home ventilation for a child. The investigators hypothesize that the intervention will increase family preparedness for decision-making and will improve clinician-family shared-decision making. Half of families will be assigned to "usual care" arm and half to the "intervention" arm. Intervention families will view the study website with study staff and will answer questions related to website content. All families will be interviewed and surveyed at 1, 6 and 12 months after enrollment. Each family will designate 1-2 physician involved in the decision about home ventilation; each physician will be interviewed and surveyed at 1 month.

DETAILED DESCRIPTION:
Across 4 centers, the investigators will recruit 150 English and/ or Spanish-speaking families (up to 2 parents per family) who are currently facing a decision about tracheostomy and home ventilation for the child. The investigators will also recruit up to 2 clinicians who are central to the decision for each child.

The first 50% of families will be assigned to "usual care" arm and the second 50% of families will be assigned to the "intervention" arm. Intervention families will view the study website with study staff and will answer questions related to website content in an interview that could last up to 2 hours. All families will be interviewed at 1, 6 and 12 months after enrollment (each interview lasts 15-30 minutes). Each family will designate 1-2 physician involved in the decision about home ventilation; each physician will be interviewed at 1 month interviews last ~15 minutes).

This is a controlled trial of a communication intervention and requires careful attention to words used. The investigators support the intention of being inclusive, and have invested considerable effort in creating a Spanish intervention and diversifying the team to include more native Spanish-speakers. However, as a communication randomized control trial (RCT), the investigators are concerned that one-off efforts to translate the website as well as using a translator, may confound the investigators interpretation of the data. Most significantly, the investigators risk not finding differences between the two arms if the investigators include those who do not speak English or Spanish.

Primary endpoints:

The investigators hypothesize that, compared to families who receive usual care related to decision-making about pediatric chronic home ventilation, families who receive the HomeVENT intervention will have increased preparedness for decision-making 1 month later.

The investigators hypothesize that, compared to families who receive usual care related to decision-making about pediatric chronic home ventilation, families who receive the HomeVENT intervention will perceive increased shared decision-making 1 month later.

The investigators hypothesize that, compared to physicians of families who receive usual care related to decision-making about pediatric chronic home ventilation, physicians of families who receive the HomeVENT intervention will perceive increased shared decision-making 1 month later.

ELIGIBILITY:
Inclusion Criteria:

1. English- or Spanish-speaking
2. Males and females; Age 18 and over.
3. Parent of a child facing a decision about home ventilation within 30 days. A "parent" will be defined as any self-identified primary caregiver (parents, grandparents, etc).

   or Physician of a child whose parents are enrolled in the study; physician must be engaged in the home ventilation decision.
4. Provision of signed and dated informed consent form (parent) or completion of oral consent (physician)
5. Stated willingness to comply with all study procedures and availability for the duration of the study
6. Access to necessary resources if choose to participate via internet or telephone

Exclusion Criteria:

1. Excluding children as they cannot be legal decision-makers
2. Non-English or Non-Spanish speaking parents, as the intervention website/ videos are only available in those two languages.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Preparedness for Decision Making among parents making decisions about home ventilation as assessed by the Preparedness for Decision Making scale. | 1 month
  The Preparedness for Decision Making scale has a possible score range of 0-100. Higher score means more prepared.
Shared Decision Making among parents making decisions about home ventilation as assessed by the CollaboRATE-Parent version scale | 1 month
  The CollaboRATE-Parent version scale is a 3 item measure. Score range 0-27. Higher score means better shared decision making.
Shared Decision Making among parents making decisions about home ventilation as assessed by the Consumer Assessment of Healthcare Providers and Systems (CAHPS-SDM) survey | 1 month
  The Consumer Assessment of Healthcare Providers and Systems scale is an 8 item measure. Score range 0-23. Higher score means better shared decision making.
Shared decision making about home ventilation for physicians as assessed by the Shared Decision Making Questionnaire - Physician (SDM-Q-DOC) version | 1 month
  The Shared Decision Making Questionnaire - Physician questionnaire is a 9 item measure. Score range 0-54. Higher score meaning better shared decision making.

SECONDARY OUTCOMES:
Change in decision making regret among parents who chose for or against home ventilation as assessed by the Decision Regret Scale | 6 months, 12 months
  The Decision Regret Scale is a 5 item scale. Score range 1-25, with higher score meaning more regret.
Change in Quality of Life expected vs. actual, among parents who faced choice about home ventilation as assessed by the Pediatric Quality of Life Family Impact Module (PEDSQL) scale | 6 months, 12 months
  The Pediatric Quality of Life Family Impact Module (PEDSQL) Score range 0-100. Higher score better quality of life.
Change in Impact of decision about home on daily life of child/ family as assessed by a qualitative interview | 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Renee Boss, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (4):
- United States (4):
  - Johns Hopkins All Childrens Hospital, Tampa, Florida
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Seattle Childrens Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Only aggregate data will be shared